CLINICAL TRIAL: NCT06241079
Title: Multi-institutional Analysis of Survival and Recurrence Patterns of Different Pathological Regression Types After Neoadjuvant Chemoradiotherapy or Radiotherapy for Esophageal Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: bc2023183
Record Dates: First submitted 2024-01-18; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ypT0N0
  Interventions: Other: non-intervention
- ypT0N+
  Interventions: Other: non-intervention
- ypT+N0
  Interventions: Other: non-intervention
- ypT+N+
  Interventions: Other: non-intervention

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
The goal of this multicenter retrospective cohort study is to evaluate the impact of different pathological regression types on survival and recurrence patterns, with a particular focus on ypT0N+ patients in patients with esophageal squamous cell carcinoma. The main questions it aims to answer are the survival and recurrence patterns among the different pathological regression types in patients with esophageal squamous cell carcinoma after neoadjuvant chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed potentially resectable ESCC, clinical stage T1-4N0-1M0 (stage I-III) according to the American Joint Committee on Cancer 6th edition staging criteria.

Exclusion Criteria:

* incomplete surgical resection, two-dimensional radiotherapy, and incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with esophageal squamous cell carcinoma (ESCC) who received NCRT or neoadjuvant radiotherapy (NRT) followed by esophagectomy from 2003 to 2022
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2003-03-31 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of surgery until the date of death from any cause or last follow-up, assessed up to 10 years.
  the time from the date of surgery to death or last follow-up (2023.01.31)